CLINICAL TRIAL: NCT03277027
Title: Health Related Lifestyle and Quality of Life in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Bo Young Hong, Assistant professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VC17OESI0046
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy; Quality of Life; Physical Activity; Physical Disability; Parenting; Sleep Disorder
Keywords: cerebral palsy; Health-Related Quality Of Life; Physical Activity
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Sleep Wake Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Non-randomized single group Accelerometer was weared for a week to check physical activity and sleep in children with cerebral palsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: interventional study — The participants wear a monitoring equipment (Actigraph) for a week. And parents do Child Health Questionnaire Parent Form 50 (CHQ-PF50), and Korean Parenting Stress Index-Short Form (K-PSI-SF)
  Other Names: Wear a monitoring equipment (Actigraph) for a week

SUMMARY:
The primary aim of this study is assessing physical activity, the quality of sleep and health related quality of life in children with cerebral palsy, and parenting stress of caregivers of the children with cerebral palsy in Korea.

DETAILED DESCRIPTION:
Monitor the physical activity, health related quality of life, parenting stress according to GMFCS level in children with cerebral palsy in Korea.

1. Physical activity and quality of sleep are monitored by wearing Actigraph for a week.
2. Health related quality of life is checked by parents withChild Health Questionnaire Parent Form 50 (CHQ-PF50).
3. Parenting stress is monitored with Korean Parenting Stress Index-Short Form (K-PSI-SF) by parents.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy, 4-19 years old

Exclusion Criteria:

* Patients with progressive brain lesions, tumors, leukodystrophies, etc.
* Children with mitochondrial myopathy
* Some diseases that are known to progress, Rett syndrome, etc.

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | Monitored for a week
  vector magnitude, steps, percentage of sedentary time monitored with Actigraph

SECONDARY OUTCOMES:
health related quality of life | Once (cross sectional)
  Checked with Child Health Questionnaire Parent Form 50 (CHQ-PF50) by parents
Parenting stress | Once (cross sectional)
  Checked with Korean Parenting Stress Index-Short Form (K-PSI-SF) by parents
Quality of sleep | Monitored for a week
  Sleep efficiency, number of awakening monitored with Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Hong, Principal Investigator — St. Vincent's hospital, The Catholic University of Korea
Locations (1):
- St. Vincent's hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD is only available to main reserchers